CLINICAL TRIAL: NCT05841719
Title: General Population Universal Capillary Screening for Chronic Autoimmune, Metabolic and Cardiovascular Diseases (UNISCREEN): Feasibility and Acceptability Pilot Study.
Brief Title: Universal Capillary Screening for Chronic Autoimmune, Metabolic and Cardiovascular Diseases: Feasibility and Acceptability Pilot Study.
Acronym: UNISCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emanuele Bosi (Other)
Collaborators: Italian Diabetes Foundation (Other)
Responsible Party: Sponsor-Investigator, Emanuele Bosi, MD, Professor of Internal Medicine, Head, General Medicine, Diabetes & Endocrinology, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UNISCREEN
Record Dates: First submitted 2023-02-03; First posted 2023-05-03 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Risk Factors; Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: capillary sampling
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population from Cantalupo, locality of the Municipality of Cerro Maggiore (MI). (Other): capillary sampling and questionnaires to test feasibility and acceptability
  Interventions: Other: Screening test

INTERVENTIONS:
Other: Screening test — Capillary blood sampling by finger-prick devices and second confirmatory venous sampling when needed.

SUMMARY:
This study represents a model for a public health program based on a general population screening for the most prevalent chronic metabolic, cardiovascular and autoimmune diseases across adulthood, childhood and adolescence. The main purpose is to assess feasibility and acceptability of using a capillary screening for this purpose. Secondly, it will be possibile to identify people at increased risk of developing one of these health conditions as well as those who are at pre-symptomatic clinical stages. Risk assessment is needed to identify prevention strategies; early diagnosis allows to start early treatment interventions aimed at reducing lifetime complications.This interventional study will enroll volunteers from Cantalupo, a locality belonging to the Municipality of Cerro Maggiore (Milan). Participants will be offered to undergo two capillary blood sampling to test blood glucose levels, glycated haemoglobin, total cholesterol, HDL-c, LDL-c, triglycerides and specific antibodies for type 1 diabetes and celiac disease. In case a participant screens positive for type I diabetes and/or celiac disease, they will be subsequently invited to undergo a new confirmatory blood draw on venous blood. Blood pressure will be also measured for each participant

DETAILED DESCRIPTION:
This is a low-risk, single-center, interventional study, assessing whether capillary screening for an early staging of the most prevalent chronic metabolic, cardiovascular and autoimmune diseases is feasible at a population-based level. The study will enroll volunteers from Cantalupo, a locality of 3095 inhabitants belonging to the Municipality of Cerro Maggiore (Milan). The main purpose is to assess feasibility and acceptability of using this public intervention. Secondary outcomes are: (i) measurement of the specific disease markers; (ii) estimation of the prevalence of the identified diseases within the population; (iii) estimation of the prevalence of the identified diseases across age classes; (iv) correlation of study disease indicators with demographics, anthropometrics and clinical data of the population , v) multiparametric risk assessment. Participants will be offered to undergo a capillary blood sampling to test blood glucose levels, glycated haemoglobin, total cholesterol , HDL-c, LDL-c, triglycerides, Glutamic Acid Decarboxylase (GADA), Insulinoma-Associated-2/Tyrosine Phosphatase (IA-2A), Insulin (IAA), Zinc Transporter-8 Autoantibodies (ZnT8A) for type I diabetes and tissue transglutaminase antibodies for celiac disease. Glucose and lipid blood levels will be detected at the time of the screening. The results of autoantibodies research for celiac disease and type 1 diabetes will be available within a few days. In case a participant screens positive for type I diabetes and/or celiac disease, they will be subsequently invited to undergo a new confirmatory blood draw on venous blood. Blood pressure will be also measured for each participant.

ELIGIBILITY:
Inclusion criteria:

* Residency in Cantalupo, locality of the Municipality of Cerro Maggiore (MI)
* Age between 1 and 100 years
* Ability to understand the purpose of the project and to sign the informed consent.

Exclusion criteria:

No exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1535 (Actual)
Dates: Start 2023-04-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
feasibility and acceptability | through study completion, an average of 1 year
  To assess feasibility and acceptability of the screening program
blood glucose and lipids level (mg/dl) | through study completion, an average of 1 year
  Capillary blood sampling will be performed by finger-prick devices.
IAA, GADA65, ZnT8, IA2 autoantibodies (U/ml) | within a few days
  Capillary blood sampling will be performed by finger-prick devices.
anti-transglutaminase autoantibodies (UA) | through study completion, an average of 1 year
  Capillary blood sampling will be performed by finger-prick devices.
systolic and diastolic blood pressure (mmHg) | through study completion, an average of 1 year
  Blood pressure measurement will be performed through a sphygmomanometer.
HbA1c (mmol/mol) | through study completion, an average of 1 year
  Glycated hemoglobin will be measured by finger-prick devices.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bosi, MD, Principal Investigator — San Raffaele Institute
Locations (1):
- Scuola dell'Infanzia Comunale Don Angelo Luzzini, Cantalupo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Ziegler AG, Hoffmann GF, Hasford J, Larsson HE, Danne T, Berner R, Penno M, Koralova A, Dunne J, Bonifacio E. Screening for asymptomatic beta-cell autoimmunity in young children. Lancet Child Adolesc Health. 2019 May;3(5):288-290. doi: 10.1016/S2352-4642(19)30028-8. Epub 2019 Feb 10. No abstract available. PMID 30745054
- [Background] Ziegler AG, Kick K, Bonifacio E, Haupt F, Hippich M, Dunstheimer D, Lang M, Laub O, Warncke K, Lange K, Assfalg R, Jolink M, Winkler C, Achenbach P; Fr1da Study Group. Yield of a Public Health Screening of Children for Islet Autoantibodies in Bavaria, Germany. JAMA. 2020 Jan 28;323(4):339-351. doi: 10.1001/jama.2019.21565. PMID 31990315
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Barry MJ, Davidson KW, Doubeni CA, Ebell M, Epling JW Jr, Herzstein J, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phipps MG, Silverstein M, Simon MA, Tseng CW. Screening for Celiac Disease: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Mar 28;317(12):1252-1257. doi: 10.1001/jama.2017.1462. PMID 28350936
- [Derived] Angiulli S, Merolla A, Borgonovo E, De Lorenzo R, Spadoni S, Fontana B, Manganaro G, Rela E, Bongiovanni A, Peracino R, Bellino C, Pata G, Bianconi E, Martinenghi S, Ulivi F, Renzi C, Bosi E; UNISCREEN Study Group. Universal capillary screening for chronic autoimmune, metabolic and cardiovascular diseases: feasibility and acceptability of the UNISCREEN study. Front Public Health. 2025 Feb 11;13:1506240. doi: 10.3389/fpubh.2025.1506240. eCollection 2025. PMID 40008147
- [Derived] Merolla A, De Lorenzo R, Ferrannini G, Renzi C, Ulivi F, Bazzigaluppi E, Lampasona V, Bosi E. Universal screening for early detection of chronic autoimmune, metabolic and cardiovascular diseases in the general population using capillary blood (UNISCREEN): low-risk interventional, single-centre, pilot study protocol. BMJ Open. 2024 Mar 5;14(3):e078983. doi: 10.1136/bmjopen-2023-078983. PMID 38448070